CLINICAL TRIAL: NCT02668900
Title: Evaluation of Decision Support for Adults Facing Implantable Cardioverter-Defibrillator Pulse Generator Replacement: A Feasibility Study
Brief Title: Decision Support for Adults Facing Implantable Cardioverter-Defibrillator Pulse Generator Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, David Birnie, MD, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UOHI-06
Record Dates: First submitted 2016-01-15; First posted 2016-01-29 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Death, Sudden, Cardiac; Death, Sudden; Cardiovascular Diseases
Keywords: Feasibility trial; Cardiovascular disease; Decision Support; Patient Decision Aid; implantable cardioverter defibrillator; implantable cardioverter defibrillator replacement
MeSH Terms: conditions — Death, Sudden, Cardiac; Death, Sudden; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision support (Experimental): The decision support intervention includes a patient decision and a decision coaching session. The patient decision aid includes a summary about the ICD's function, and the risks and benefits (including probabilities) associated with the option of replacing or not replacing the ICD. The decision coaching session will be led by a trained, non-directive decision coach who will provide support that aims to develop patients' skills in thinking about the options, assess their values associated with each option, and prepare them to discuss the decision in a consultation with their physician. The final decision, whether to replace or not replace the ICD, will be made with their treating physician (e.g., cardiologist, electrophysiologist).
  Interventions: Behavioral: Decision Support
- Usual care (No Intervention): The control group will not receive the decision support intervention prior to consultation with the physician.

INTERVENTIONS:
Behavioral: Decision Support — The decision support intervention includes a patient decision and a decision coaching session. The patient decision aid includes a summary about the ICD's function, and the risks and benefits (including probabilities) associated with the option of replacing or not replacing the ICD. The decision coaching session will be led by a trained, non-directive decision coach who will provide support that aims to develop patients' skills in thinking about the options, assess their values associated with each option, and prepare them to discuss the decision in a consultation with their physician. The final decision, whether to replace or not replace the ICD, will be made with their treating physician (e.g., cardiologist, electrophysiologist).
  Arms: Decision support

SUMMARY:
The implantable-cardioverter defibrillator (ICD) is a small medical device used to treat dangerously fast and potentially life-threatening heart rates. For patients at risk, the ICD can detect an abnormal rhythm and provide life-saving therapy by delivering a shock. ICD therapy has risks and benefits that should be weighed from each patient's perspective. An ICD battery needs to be surgically replaced 4 to 7 years to ensure ongoing function. At present, the majority of these batteries are automatically changed without eliciting patients' preferences. There is a need for a better way to engage with patients. Patients want to be involved in their healthcare decisions, yet more than half of patients with an ICD do not know that ICD replacement is optional. To ensure that patients are receiving treatment that they value and want, members of the interprofessional team should ensure that treatment decisions align with patients' expectations, values and preferences. This rests on the principle of shared decision making in which members of the healthcare team and patients deliberate together to arrive at a decision which best reflects the preferences and values of the patient. To facilitate the achievement of this goal, a patient decision aid (PDA) can be used. As a result, the investigators developed PDA for ICD replacement. The purpose of this feasibility trial is to collect preliminary data to test the feasibility of conducting a larger trial, and to evaluate the PDA for its acceptability and ease of use. Eligible and consented participants facing ICD replacement will be randomized to receive the decision aid or to usual care. The investigators will assess if this decision aid can improve participants' knowledge on ICD therapy and the replacement surgery, increase patients' perceived involvement in the decision, and determine whether their actual choice reflects their personal values.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) due to a ventricular arrhythmia is a serious cause of cardiovascular death in Canada. The implantable cardioverter defibrillator (ICD) can reduce the incidence of SCD in high-risk patients by delivering an internal shock to restore a normal rhythm. The life expectancy of an ICD generator is estimated between four and seven years, and must be surgically replaced to ensure ongoing function. Implantable cardioverter-defibrillator (ICD) replacement is becoming increasingly common constituting nearly 40% of all ICD procedures. For the most part, ICDs are automatically replaced. With every ICD replacement, the net benefit of continued ICD therapy should be assessed individually in view of the procedural risks, inappropriate shocks, psychological risks, changes in health status, and the potential for harm and suffering at end-of-life. Some studies have shown that the mortality benefit of an ICD attenuates with advancing age and comorbidities.

There are many legitimate reasons for declining ICD generator replacement. The chronic nature of a cardiac condition and/or the diagnosis of a life-limiting disease since initial implantation may compel a patient to reconsider their health care goals from supporting quantity of life, to prioritizing one of quality. This is an important distinction as the ICD can prolong the dying process by delivering shock(s) which can result in pain and discomfort for the patient, and helplessness for witnesses. Other patients have reported psychological distress, while others report only truly understanding the effects of living with an ICD after receiving one, possibly leading to changes in treatment preference when they are faced with the decision to replace. Also, the replacement procedure includes a substantially greater risk for infection and reoperation as compared to the initial implantation.

These complexities warrant decision support to prepare patients to make decisions. Yet, no means exists to support patients' decision-making in the context of ICD replacement. A decision support intervention (including a patient decision aid with decision coaching) was developed using a user-centered design with various stakeholders and potential end-users, which could moderate treatment related uncertainty and prepare patients to make high quality decisions that are informed and based on their personal preferences and values.

Objectives:

1. Conduct a pilot randomized controlled trial (RCT) to determine the feasibility of conducting a larger trial.
2. To determine the effect of the decision support intervention for adults faced with ICD replacement on attributes of decision quality and decision-making processes

ELIGIBILITY:
Inclusion Criteria:

* ICD battery nearing depletion or at elective replacement indicator
* Able to speak and read in English
* Able to provide informed consent; or if incapable of providing informed consent, can be obtained by the patient's appointed substitute decision-maker or power of attorney for personal care.

Exclusion Criteria:

* Participants and/or substitute decision maker unable to understand the patient decision aid or decision coaching session due to language barrier or visual impairment
* Participants with cardiac resynchronization therapy (CRT) or participants eligible for an upgrade to CRT.
* Participants with conduction system disease who are pacemaker dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Pilot RCT (feasibility measure): Participant referral/recruitment rate. | Baseline to 6 months
  In this feasibility RCT, the feasibility regarding key processes to the success of a larger trial will be assessed. The investigators will descriptively collect the proportion of participant referral versus recruitment rate.
Pilot RCT (feasibility measure): Completion of decision support intervention | Baseline to 6 months
  In this feasibility RCT, the feasibility regarding key processes to the success of a larger trial will be assessed. The investigators will descriptively collect the rate of participants who complete the decision support intervention.
PIlot RCT (feasibility measure) | Baseline to 6 months
  In this feasibility RCT, the feasibility regarding key processes to the success of a larger trial will be assessed. The investigators will descriptively collect the proportion of missing data from the questionnaires.

SECONDARY OUTCOMES:
Knowledge | 1 month; intervention and usual care groups
  The investigators developed a knowledge test based on the content of the patient decision aid. It was endorsed for validity by the patient decision aid (PtDA) development team using a standardized template in the form of true or false questions. There are six questions meant to assess a patient's understanding of their heart condition, treatment options, and risks and benefits of each option. Correct answers will be summed to determine an overall score.
Decisional conflict | 1 month, 6 months, 12 months post; intervention and usual care groups
  The Decisional Conflict Scale measures a person's perception of the difficulty in making a decision, the extent to which they feel uncertain about treatment options, are knowledgeable about the risks and benefits of options, clear about personal values, and supported in decision making. The scale has good test-retest reliability (Cronbach's alpha coefficients > 0.78) and predictive validity.
Values about ICD replacement | 1 month; intervention and usual care groups
  The investigators developed a values clarification exercise based on the characteristics of the ICD replacement decision. It was endorsed for validity by the patient decision aid (PtDA) development team using a standardized template in the form of likert-type questions. There are four statements meant to help participants consider the risks and benefits of replacing or not replacing the ICD battery than matter most to them. There are no right or wrong answers.
Preferred option | Baseline visit, 1 month, 6 months, 12 months; intervention and usual care groups
  Preferred option will be measured by asking patients whether they prefer to have their ICD's pulse generator replaced, not replaced, or whether they are unsure using the 15-point Choice Predisposition Scale that demonstrates a patient's inclination toward a given option. This scale has a test-retest coefficient >0.90.
Perceptions of involvement in decision-making | 6 months, 12 months; intervention and usual care groups
  This will be measured using a modified version of Strull, Lo, & Charles's (1984) role in decision-making survey. Five statements rest along the continuum of how decisions can be made between patients and providers. Participants must select the statement that best represents their perceived involvement in the final decision
The Medical Outcomes Trust Short Form (SF-36v2) | Baseline visit intervention and usual care groups
  The SF-36 is a reliable and valid generic health related quality of life scale (HRQL) comprised of 36 items. Associations between HRQL and decision choice will be made.
Acceptability and Usability of Decision Support | 1 month; intervention group only
  Intervention group participants will be asked common acceptability and usability questions extensively used for evaluating PtDAs during development (Barry, Cherkin, Chang, Fowler, & Skates, 1997; Kushniruk & Patel, 2004; O'Connor & Cranney, 2002). Patients' satisfaction with decision coaching will be measured using the Genetic Counseling Satisfaction Scale and perceptions of decision coach neutrality (Schwalm, Stacey, Pericak, & Natarajan, 2012; Tercyak, Johnson, Roberts, & Cruz, 2001). This scale has face validity and a reliability coefficient of alpha 0.80 to 0.90 in genetic counselling contexts with adults.

OTHER OUTCOMES:
Actual choice | 6 months, 12 months; intervention and usual care groups
  The number of participants who choose to accept ICD replacement, decline ICD replacement, or defer their decision to later.
Survival | 6 months, 12 months; intervention and usual care groups
  The number of participants who are alive or dead at 6 months. If participant is dead, include cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Stacey, RN, PhD, Study Director — University of Ottawa; Ottawa Hospital Research Institute
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewis KB, Birnie D, Carroll SL, Brousseau-Whaley C, Clark L, Green M, Nair GM, Nery PB, Redpath C, Stacey D. Decision Support for Implantable Cardioverter-Defibrillator Replacement: A Pilot Feasibility Randomized Controlled Trial. J Cardiovasc Nurs. 2021 Mar-Apr 01;36(2):143-150. doi: 10.1097/JCN.0000000000000694. PMID 32453274